CLINICAL TRIAL: NCT05859802
Title: Effects of Physical Therapy and Dalfampridine on Functional Mobility and Lower Extremity Strength in Non Ambulatory Persons With Multiple Sclerosis
Brief Title: Effects of Physical Therapy and Dalfampridine on Functional Mobility in Non Ambulatory Persons With Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: D'Youville College (Other)
Collaborators: Acorda Therapeutics (Industry); University at Buffalo (Other)
Responsible Party: Principal Investigator, Lacey Bromley, Project Manager, D'Youville College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RMD0690511A
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: Dalfampridine; Functional Mobility; Non ambulatory; Cognition; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were blinded and randomized into 2 groups; Group 1 received physical therapy for 12 weeks while taking Dalfampradine 10 mg two times day and Group 2 received physical therapy while taking a placebo pill two times a day.
  Both investigators that were preforming the testing and treatment were blinded as to subject group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Group (Experimental)
  Interventions: Drug: Dalfampridine Pill
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine Pill — Subjects were blinded and randomized into 2 groups; Group 1 received physical therapy 2 x a week for 12 weeks while taking dalfampridine 10 mg two times day
  Other Names: Physical Therapy
  Arms: Drug Group
Drug: Placebo — Subjects were blinded and randomized into 2 groups; Group 1 received physical therapy 2 x a week for 12 weeks while taking a placebo pill two times day
  Arms: Placebo Group

SUMMARY:
The goal of this interventional double blind, randomized placebo controlled trial was to assess the change in functional mobility, quality of life and cognition for subjects who receive physical therapy and take dalfampridine vs those who receive physical therapy and take a placebo in non ambulatory persons with multiple sclerosis. The main question[s] it aims to answer are:

1. Does the addition of dalfampridine to Physical Therapy improve functional outcomes compared to Physical Therapy alone
2. Does Physical Therapy improve functional outcomes in patients who are non ambulatory

DETAILED DESCRIPTION:
This randomized control trial examined the effectiveness of dalfampridine when administered in conjunction with 12 weeks of physical therapy compared to physical therapy and a placebo on function, quality of life (QoL) and cognition in non-ambulatory pwMS.

Specific Aim 1: Assess the change in standing tolerance, transfers, repeated sit to stand, QoL and cognitive processing for non-ambulatory individuals with MS between subjects on Dalfampridine who receive physical therapy and those who participate in physical therapy and receive a placebo. Enhancing the propagation of action potentials along axons in addition to regularly contracting the muscles through exercise may have a greater effect on strength and functional mobility.

Specific Aim 2: Assess the functional, strength and cognitive changes within all subjects receiving PT 2x a week for 12 weeks. Evidence supporting the effectiveness of physical therapy in this population is extremely limited.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older confirmed MS diagnosis
* Expanded Disability Status Scale (EDSS) of 7.0 or higher
* No steroid treatment in the last 30 days or a relapse in the last 90 days, and MS considered stable
* Capable of performing requirements of Physical Therapy (PT) treatment including at least a 2/5 manual muscle test in 50% or more of the major muscle groups

Exclusion Criteria:

* History of seizure disorder
* Major cognitive or mental illness that prevented their ability to provide consent
* Evidence of other medical cause of cognitive impairment besides MS
* Severe joint contractures that limited the patients ability to move within full active range of motion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07-13 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2016-01-09 (Actual)

PRIMARY OUTCOMES:
MSQOL -54 | Baseline
MSQOL -54 | 6 weeks
MSQOL -54 | 12 weeks
Five time Sit to Stand | Baseline
Five time Sit to Stand | 6 weeks
Five time Sit to Stand | 12 weeks

SECONDARY OUTCOMES:
Symbol Digit Modalities Test | Baseline
Symbol Digit Modalities Test | 6 weeks
Symbol Digit Modalities Test | 12 weeks
Wheel chair to Mat transfers - Functional Independence Measure | Baseline
Wheel chair to Mat transfers - Functional Independence Measure | 6 weeks
Wheel chair to Mat transfers - Functional Independence Measure | 12 weeks
Standing Tolerance | Baseline
  Standardized performance of static standing has not been published. For this study the subject will be positioned with the wheelchair directly in front of a sink counter. The examiner will ask the patient to stand up facing the sink counter, keeping two hands on the counter [at the sink cutout area]. The examiner will stand next to the subject and guard as needed during this task. Upon standing upright the examiner will start the stopwatch. The time will be stopped when the subject is unable to maintain an upright posture defined as flexing of the hips and knees or bending the trunk forward to lean on the counter. Two trials will be performed (separated by a 2 minute rest) with the longest time in upright standing recorded.
Standing Tolerance | 6 weeks
  Standardized performance of static standing has not been published. For this study the subject will be positioned with the wheelchair directly in front of a sink counter. The examiner will ask the patient to stand up facing the sink counter, keeping two hands on the counter [at the sink cutout area]. The examiner will stand next to the subject and guard as needed during this task. Upon standing upright the examiner will start the stopwatch. The time will be stopped when the subject is unable to maintain an upright posture defined as flexing of the hips and knees or bending the trunk forward to lean on the counter. Two trials will be performed (separated by a 2 minute rest) with the longest time in upright standing recorded.
Standing Tolerance | 12 weeks
  Standardized performance of static standing has not been published. For this study the subject will be positioned with the wheelchair directly in front of a sink counter. The examiner will ask the patient to stand up facing the sink counter, keeping two hands on the counter [at the sink cutout area]. The examiner will stand next to the subject and guard as needed during this task. Upon standing upright the examiner will start the stopwatch. The time will be stopped when the subject is unable to maintain an upright posture defined as flexing of the hips and knees or bending the trunk forward to lean on the counter. Two trials will be performed (separated by a 2 minute rest) with the longest time in upright standing recorded.
9 Hole Peg Test | Baseline
9 Hole Peg Test | 6 weeks
9 Hole Peg Test | 12 weeks

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-06-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT05859802/Prot_SAP_000.pdf
  • Informed Consent Form (2011-07-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT05859802/ICF_001.pdf